CLINICAL TRIAL: NCT00186901
Title: Diminished Bone Mineral Density in Survivors of Childhood Acute Lymphoblastic Leukemia (ALL): A Severity-Adapted Clinical Trial
Brief Title: A Severity-Adapted Clinical Trial of Diminished Bone Mineral Density in Acute Lymphoblastic Leukemia Survivors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BONEII
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2012-03-27 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2011-12

CONDITIONS: Leukemia, Lymphoblastic, Acute; Osteoporosis
Keywords: Bone Density
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Osteoporosis | interventions — Calcium Carbonate; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1A (Placebo Comparator): Nutritional counseling + placebo
  Interventions: Other: Placebo
- 1B (Experimental): Nutritional counseling + supplementation with calcium, 1000mg/day + vitamin D, 800 units/day, for a 2 year period
  Interventions: Drug: Calcium carbonate (Tums), vitamin D

INTERVENTIONS:
Drug: Calcium carbonate (Tums), vitamin D — Calcium carbonate 100mg/day (Tums), vitamin D 800 units/day
  Arms: 1B
Other: Placebo — Placebo
  Arms: 1A

SUMMARY:
Research studies have shown that children who are long-term survivors of childhood leukemia may be at greater risk for early bone loss called osteoporosis. This bone loss may lead to a greater risk of broken bones and other spine and bone problems. However, researchers still do not know much about how frequently this long-term side effect may occur and how severe the problem is.

St. Jude Children's Research Hospital researchers want to determine the frequency and severity of this side effect. They are also studying whether taking calcium and Vitamin D supplements can help children at risk for osteoporosis and if certain factors can be identified -- such as age at diagnosis, cancer treatments, or family history -- that may increase the chances of having osteoporosis. Researchers will take an x-ray study called quantitative computed tomography (QCT) to measure bone mineral density (BMD). The BMD is a measure of bone strength. If a subject's BMD falls below the average, he/she will be assigned to one of two groups. Subjects will be randomly assigned (like tossing a coin) to receive calcium and vitamin D pills. The other half will receive placebo pills that look like the calcium and vitamin D pills.

DETAILED DESCRIPTION:
The main objectives of the study are:

* To estimate, using quantitative computed tomography (QCT), the prevalence of diminished bone mineral density (BMD) in patients treated with contemporary, protocol-based multiagent chemotherapy (+cranial irradiation) for childhood acute lymphoblastic leukemia (ALL).
* To investigate possible risk factors for the development of diminished BMD in patients treated with contemporary protocol-based therapy for childhood ALL. Factors to be examined include patient characteristics (age at the time of treatment, gender, race, body mass index, physical activity and nutritional status, menarchal status, oral contraceptive use, growth hormone therapy, smoking and alcohol intake, birth weight, fracture history); treatment effects (intensity of treatment with antimetabolites and glucocorticoids; history of cranial irradiation); and genetic predisposition (i.e., vitamin D and CYP3A4 receptor polymorphism and family history of osteoporosis).
* To evaluate, in a prospective placebo-controlled double-blinded randomized trial, the effects of vitamin D and calcium supplementation in addition to nutritional counseling on BMD in patients with BMD scores below the mean for age- and gender-matched controls, compared to an educational program of nutritional counseling alone.

Secondary Aim

* To evaluate, in a prospective randomized trial, the correlation between BMD as determined by QCT and BMD as determined by dual energy x-ray absorptiometry (DEXA) in patients with BMD more than one standard deviation (SD) below the mean for age- and gender-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a survivor of acute lymphoblastic leukemia.
* Patient was treated on St. Jude Children's Research Hospital's Total XI, XII, or XIII treatment protocol.
* Patient is at least five years out from completion of therapy and is in first remission

Exclusion Criteria:

* Active disease
* Pregnant or lactating females
* Inability to chew and swallow pills
* Currently taking more than 800 mg supplemental calcium or 800 IU vitamin D
* Anemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2000-07; Primary Completion 2009-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue C. Kaste, D.O., Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Metabolic Bone Center at the University of Tennessee, Memphis, Tennessee
  - Preventive Medicine, University of Tennessee, Memphis, Tennessee

REFERENCES:
- [Background] Kaste SC, Rai SN, Fleming K, McCammon EA, Tylavsky FA, Danish RK, Rose SR, Sitter CD, Pui CH, Hudson MM. Changes in bone mineral density in survivors of childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2006 Jan;46(1):77-87. doi: 10.1002/pbc.20553. PMID 16106430
- [Background] Crom DB, Tyc VL, Rai SN, Deng X, Hudson MM, Booth A, Rodrigues LN, Zhang L, McCammon E, Kaste SC. Retention of survivors of acute lymphoblastic leukemia in a longitudinal study of bone mineral density. J Child Health Care. 2006 Dec;10(4):337-50. doi: 10.1177/1367493506067886. PMID 17101625
- See also: St. Jude Children's Research Hospital — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 429 patients were recruited at St. Jude Children's Research Hospital between August 7, 2000 and July 27, 2006. 4 patients were found to be ineligible and 1 patient was taken off study per the PI's request. 424 patients were available at baseline.
Pre-assignment Details: 424 total patients were enrolled on the study. 149 patients were ineligible for randomization. 275 patients were identified with Bone Mineral Density (BMD) Z-scores > 0 and thus were eligible for intervention and were randomized to receive either Calcium and Vitamin D supplementation or placebo.
Groups:
- Placebo Group: Nutritional counseling + placebo
- Supplement Group: Nutritional counseling + supplementation with calcium, 1000mg/day + vitamin D, 800 units/day, for a 2 year period
- Patients Ineligible for Randomization: 424 patients were enrolled into the study, 149 were ineligible for randomization.
Period: Overall Study
Arm/Group | Placebo Group | Supplement Group | Patients Ineligible for Randomization
Started | 134 | 141 | 149
Baseline | 134 | 141 | 0
12 Month Follow-up | 117 | 122 | 0
24 Month Follow-up | 106 | 107 | 0
Completed | 85 | 96 | 0
Not Completed | 49 | 45 | 149
Not completed — Pregnancy | 6 | 3 | 0
Not completed — Lost to Follow-up | 6 | 3 | 0
Not completed — Bone Mineral Density dropped > 5% | 9 | 7 | 0
Not completed — ALL relapse or second malignancy | 1 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 0
Not completed — Open label | 3 | 2 | 0
Not completed — Limited adherence to study requirements | 20 | 23 | 0
Not completed — Bone Mineral Density > 0 | 0 | 0 | 149

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Supplement Group | Patients Ineligible for Randomization | Total
Number analyzed (Participants) | 134 | 141 | 149 | 424
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.9 (5.6) | 17.6 (6.3) | 19.2 (6.6) | 17.8 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 63 | 87 | 206
  Male | 78 | 78 | 62 | 218

OUTCOME MEASURES:

1. Primary Outcome: Effect of Taking Calcium and Vitamin D Supplements on Bone Mineral Density (BMD)
Description: The effect of taking calcium and vitamin D supplements was measured using Quantitative Computed Tomography (QCT) to calculate a QTC Z score. A standardized Z-score was calculated to indicate the difference between the patient's Bone Mineral Density (BMD) and the mean value for age and gender-appropriate controls. Z-scores from 0 to +2 are considered normal, above +2 are considered to be elevated, from 0 to -1 are considered to represent a mild BMD deficit, between -1 and -2 are considered to represent moderate deficits, and below -2 are considered to represent severe deficits.
Time Frame: Baseline, 12 months, 24 months, and at 36 months or study end
Population: Of the 275 pts identified with BMD z-scores < 0, 134 were randomized to the placebo group and 141 to the supplement group. Bone Mineral Density QCT Z-scores were calculated at baseline, 12 months, 24 months, and at 36 months or study end.
Measure: Median (Full Range); unit: Z-Score
Groups:
- Placebo: Placebo Group (Placebo Comparator 1A): Patients who received placebo pills.
- Supplement: CVD Supplement Group (Experimental 1B): Patients who received calcium and vitamin D supplementation.
Arm/Group | Placebo | Supplement
Number analyzed (Participants) | 134 | 141
Z-Score
  Baseline | -0.95 [-3.09 to -0.05] | -0.97 [-3.94 to -0.04]
  12 Months | -0.87 [-3.23 to 0.85] | -1.04 [-4.32 to 0.58]
  24 Months | -0.72 [-2.61 to 0.91] | -0.76 [-3.75 to 1.23]
  36 Months (study end) | -0.56 [-2.96 to 1.36] | -0.61 [-4.23 to 2.02]
Statistical Analysis 1: Comparison: Placebo vs Supplement; Baseline where N=134; Test type: Superiority or Other; p = 0.86, Wilcoxon Test; Median Difference (Final Values) = -0.02
Statistical Analysis 2: Comparison: Placebo vs Supplement; 12 Month BMD Z-Score Calculation where N=109; Test type: Superiority or Other; p = 0.99, Wilcoxon Test; Median Difference (Final Values) = -0.17
Statistical Analysis 3: Comparison: Placebo vs Supplement; 24 Month BMD Z-Score calculation where N=91; Test type: Superiority or Other; p = 0.54, Wilcoxon Test; Median Difference (Final Values) = -0.04
Statistical Analysis 4: Comparison: Placebo vs Supplement; 36 Month (End of Study) BMD Z-Score calculation where N=84; Test type: Superiority or Other; p = 0.31, Wilcoxon Test; Median Difference (Final Values) = -0.04

2. Primary Outcome: Bone Mineral Density in Male and Female ALL Survivors
Description: Using bone mineral density Z-score, assess relationship between predisposing factors (gender) and bone mineral density; a negative value indicates a deficit in bone mineral density.
Time Frame: Baseline
Population: Baseline participants were assessed to determine whether gender was a pre-disposing factor for bone mineral density.
Measure: Median (Standard Error); unit: Z-score
Groups:
- Male: 218 males were eligible for the study
- Female: 206 females were eligible for the study
Arm/Group | Male | Female
Number analyzed (Participants) | 218 | 206
Z-score | -0.62 (1.18) | -0.3 (1.18)
Statistical Analysis 1: Comparison: Male vs Female; Test type: Superiority or Other; p = 0.0004, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.32

3. Primary Outcome: Bone Mineral Density by Race of ALL Survivors
Description: Using bone mineral density Z-score, assess relationship between predisposing factors (race) and bone mineral density; a negative value indicates a deficit in bone mineral density.
Time Frame: Baseline
Population: Assess baseline participants to determine whether race contributed to bone mineral density.
Measure: Median (Standard Error); unit: Z-score
Groups:
- White: 365 white patients were eligible for the study
- Non-white: 59 non-white were eligible for the study
Arm/Group | White | Non-white
Number analyzed (Participants) | 365 | 59
Z-score | -0.54 (1.14) | 0.15 (1.56)
Statistical Analysis 1: Comparison: White vs Non-white; Test type: Superiority or Other; p = 0.0023, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.69

4. Primary Outcome: Bone Mineral Density by Age Group of ALL Survivors
Description: Using bone mineral density Z-score, assess relationship between predisposing factors (age groups) and bone mineral density; a negative value indicates a deficit in bone mineral density.
Time Frame: Baseline
Population: Assess baseline participants to determine whether age was a contributing factor in bone mineral density.
Measure: Median (Standard Error); unit: Z-score
Groups:
- 9 to 13 Years: 98 patients between the ages of 9 and 13 were eligible for the study
- 13 to 18 Years: 139 patients between the ages of 13 and 18 were eligible for the study
- 18 to 22 Years: 74 patients between the ages of 18 and 22 were eligible for the study
- Above 22 Years: 113 patients greater than 22 years of age were eligible for the study
Arm/Group | 9 to 13 Years | 13 to 18 Years | 18 to 22 Years | Above 22 Years
Number analyzed (Participants) | 98 | 139 | 74 | 113
Z-score | -0.6 (1.1) | -0.54 (1.21) | -0.59 (1.2) | -0.25 (1.29)
Statistical Analysis 1: Comparison: 9 to 13 Years vs 13 to 18 Years vs 18 to 22 Years vs Above 22 Years; Test type: Superiority or Other; p = 0.0092, Kruskal-Wallis

5. Secondary Outcome: Quantitative Computed Tomography (QCT) and Dual Energy X-ray Absorptiometry (DXA) Scan Scores for Bone Mineral Density.
Description: To compare the bone mineral density scores determined by Quantitative Computed Tomography (QCT) with those determined by dual energy x-ray absorptiometry (DXA) scan. 121 patients at baseline were assessed by both method the QCT and DXA methods to assess Bone Mineral Density.
Time Frame: Baseline
Population: 275 patients were assessed at baseline and received a QCT Scan. 121 patients were also assessed using the DEXA Scan. Comparison of the two methods used 121 paired studies to arrive at a correlation coefficient.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Placebo - (QCT): 134 patients were assessed at baseline using the QCT scan.
- Placebo - (DXA): 60 of the 134 baseline patients also had a DXA scan.
- Supplement - (QCT): 141 patients were assessed at baseline using the QCT scan.
- Supplement - (DXA): 61 of the 141 baseline patients also had a DXA scan.
Arm/Group | Placebo - (QCT) | Placebo - (DXA) | Supplement - (QCT) | Supplement - (DXA)
Number analyzed (Participants) | 134 | 60 | 141 | 61
Z-score | -1.06 (0.70) [0.25 to 0.55] | -1.30 (1.21) | -1.09 (0.74) | -1.18 (1.02)
Statistical Analysis 1: Comparison: Placebo - (QCT) vs Placebo - (DXA) vs Supplement - (QCT) vs Supplement - (DXA); 275 received a QCT and 121 received a DXA scan. 121 paired scans were evaluated; Test type: Superiority or Other; p < 0.0001, Z-test; Correlation coefficient = 0.41, 95% CI 2-sided [0.25 to 0.55]

6. Secondary Outcome: Quantitative Computed Tomography (QCT) and Dual Energy X-ray Absorptiometry (DXA) Scan Scores for Bone Mineral Density.
Description: To compare the bone mineral density scores determined by Quantitative Computed Tomography (QCT) with those determined by dual energy x-ray absorptiometry (DXA) scan. 218 patients were assessed at 12 months for QCT. 94 were evaluated using DXA. 94 patients received both scans.
Time Frame: 12 months
Population: 218 patients were assessed at the 12 months interval and received a QCT Scan. 94 patients were also assessed using the DXA Scan. Comparison of the two methods used 94 paired studies to arrive at a correlation.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Placebo - (QCT); Supplement - (QCT): 109 patients were assessed at 12 months using the QCT scan.
- Placebo - (DXA); Supplement - (DXA): 47 of the 109 patients assessed at 12 months also had a DXA scan.
Arm/Group | Placebo - (QCT) | Placebo - (DXA) | Supplement - (QCT) | Supplement - (DXA)
Number analyzed (Participants) | 109 | 47 | 109 | 47
Z-score | -1.02 (0.87) [0.38 to 0.67] | -1.20 (1.36) | -1.04 (0.89) | -0.79 (0.93)
Statistical Analysis 1: Comparison: Placebo - (QCT) vs Placebo - (DXA) vs Supplement - (QCT) vs Supplement - (DXA); 218 patients were assessed at 12 months and received a QCT Scan. 94 patients were also assessed using the DEXA Scan. Comparison of the two methods used 94 paired studies to arrive at a correlation coefficient; Test type: Superiority or Other; p < 0.0001, Z-test; Correlation coefficient = 0.54, 95% CI 2-sided [0.38 to 0.67]

7. Secondary Outcome: Quantitative Computed Tomography (QCT) and Dual Energy X-ray Absorptiometry (DXA) Scan Scores for Bone Mineral Density.
Description: To compare the bone mineral density scores determined by Quantitative Computed Tomography (QCT) with those determined by dual energy x-ray absorptiometry (DXA) scan. 188 patients were assessed at 24 months by the QCT method and 90 were evaluated using the DXA methods to assess Bone Mineral Density. 90 patients received both scans.
Time Frame: 24 months
Population: 188 patients were assessed at the 24 months interval and received a QCT Scan. 90 patients were also assessed using the DXA Scan. Comparison of the two methods used 90 paired studies to arrive at a correlation.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Placebo - (QCT): 91 patients were assessed at 24 months using the QCT scan.
- Placebo - (DXA): 39 of the 91 patients assessed at 24 months also had a DXA scan.
- Supplement - (QCT): 97 patients were assessed at 24 months using the QCT scan.
- Supplement - (DXA): 51 of the 97 patients assessed at 24 months also had a DXA scan.
Arm/Group | Placebo - (QCT) | Placebo - (DXA) | Supplement - (QCT) | Supplement - (DXA)
Number analyzed (Participants) | 91 | 39 | 97 | 51
Z-score | -0.75 (0.82) [0.36 to 0.66] | -0.77 (1.31) | -0.84 (0.86) | -0.60 (1.07)
Statistical Analysis 1: Comparison: Placebo - (QCT) vs Placebo - (DXA) vs Supplement - (QCT) vs Supplement - (DXA); 188 patients were assessed at baseline and received a QCT Scan. 90 patients were also assessed using the DEXA Scan. Comparison of the two methods used 90 paired studies to arrive at a correlation coefficient; Test type: Superiority or Other; p < 0.0001, Z-test; Correlation coefficient = 0.53, 95% CI 2-sided [0.36 to 0.66]

8. Secondary Outcome: Quantitative Computed Tomography (QCT) and Dual Energy X-ray Absorptiometry (DXA) Scan Scores for Bone Mineral Density.
Description: To compare the bone mineral density scores determined by Quantitative Computed Tomography (QCT) with those determined by dual energy x-ray absorptiometry (DXA) scan. 180 patients were assessed at 36 months by the QCT method and 89 were evaluated using the DXA methods to assess Bone Mineral Density. 89 patients received both scans.
Time Frame: 36 months
Population: 180 patients were assessed at the 36 months interval and received a QCT Scan. 89 patients were also assessed using the DEXA Scan. Comparison of the two methods produced 89 paired studies to arrive at a correlation.
Measure: Median (Standard Deviation); unit: Z-score
Groups:
- Placebo - (QCT): 84 patients were assessed at 36 months using the QCT scan.
- Placebo - (DXA): 36 of the 84 patients assessed at 36 months also had a DXA scan.
- Supplement - (QCT): 96 patients were assessed at 36 months using the QCT scan.
- Supplement - (DXA): 53 of the 96 patients assessed at 36 months also had a DXA scan.
Arm/Group | Placebo - (QCT) | Placebo - (DXA) | Supplement - (QCT) | Supplement - (DXA)
Number analyzed (Participants) | 84 | 36 | 96 | 53
Z-score | -0.54 (0.86) [0.3 to 0.63] | -0.63 (1.14) | -0.71 (0.98) | -0.63 (1.00)
Statistical Analysis 1: Comparison: Placebo - (QCT) vs Placebo - (DXA) vs Supplement - (QCT) vs Supplement - (DXA); 180 patients were assessed at 36 months and received a QCT Scan. 89 patients were also assessed using the DXA Scan. Comparison of the two methods used 89 paired studies to arrive at a correlation coefficient; Test type: Superiority or Other; p < 0.0001, Z-test; Correlation coefficient = 0.48, 95% CI 2-sided [0.30 to 0.63]

9. Secondary Outcome: Mean QCT Z-Score by Apa1 Vitamin D Receptor Genotype
Description: The Apa1 Vitamin D Receptor has been associated with bone mineral density and bone turnover markers in various patient cohorts but has not been investigated I survivors of childhood
Time Frame: At enrollment
Population: Of the 424 patients screened, 417 participants consented for genetic testing. Of the 417 patients screened for the Apa 1 vitamin D receptor, only 68 had the AA genotype, 104 had the Aa genotype, and 49 had the aa genotype.
Measure: Mean (Standard Deviation); unit: QCT Z-Score
Groups:
- Apa 1 - AA Genotype: The AA genotype was observed in 68 (16.31%) out of 417 participants, with a median BMD Z score (a unit-less measure comparing to the age and gender matched national average) of -0.56.
- Apa 1 - Aa Genotype: The Aa genotype was observed in 104 (24.94%) out of 417 participants, with a median BMD Z score of -0.44.
- Apa 1 - aa Genotype: The aa genotype was present in 49 (11.75%) out of 417 participants, with a median BMD Z score of -0.57.
Arm/Group | Apa 1 - AA Genotype | Apa 1 - Aa Genotype | Apa 1 - aa Genotype
Number analyzed (Participants) | 68 | 104 | 49
QCT Z-Score | -0.56 (1.27) | -0.44 (1.28) | -0.57 (1.13)
Statistical Analysis 1: Comparison: Apa 1 - AA Genotype vs Apa 1 - Aa Genotype vs Apa 1 - aa Genotype; Test type: Superiority or Other; p = 0.40, Kruskal Wallis

10. Secondary Outcome: Mean QCT Z-Score by Bsm 1 Vitamin D Receptor Genotype
Description: The Bsm1 Vitamin D Receptor has been associated with bone mineral density and bone turnover markers in various patient cohorts but has not been investigated I survivors of childhood
Time Frame: At enrollment
Population: Of the 424 patients screened, 417 participants consented for genetic testing. Of the 417 patients screened for the Bsm 1 vitamin D receptor, only 41 had the BB genotype, 65 had the Bb genotype, and 77 had the bb genotype.
Measure: Mean (Standard Deviation); unit: QCT Z-Score
Groups:
- Bsm - BB Genotype: The BB genotype was observed in 41 (09.83%) out of 417 participants, with a median BMD Z score (a unit-less measure comparing to the age and gender matched national average) of -0.5.
- Bsm - Bb Genotype: The Bb genotype was observed in 65 (15.59%) out of 417 participants, with a median BMD Z score of -0.17.
- Bsm - bb Genotype: The bb genotype was observed in 77 (18.47%) out of 417 participants, with a median BMD Z score of -0.17.
Arm/Group | Bsm - BB Genotype | Bsm - Bb Genotype | Bsm - bb Genotype
Number analyzed (Participants) | 41 | 65 | 77
QCT Z-Score | -0.5 (1.2) | -0.17 (1.25) | -0.17 (1.24)
Statistical Analysis 1: Comparison: Bsm - BB Genotype vs Bsm - Bb Genotype vs Bsm - bb Genotype; Test type: Superiority or Other; p = 0.21, Kruskal Wallis

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events from August, 2000 through July, 2006.
Arm/Group | Placebo Group | Supplement Group | Patients Ineligible for Randomization
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/141 | 0/149
Other Adverse Events (participants affected / at risk) | 0/134 | 0/141 | 0/149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes